CLINICAL TRIAL: NCT02525809
Title: Incidence of Dual Mobility Polyethylene Wear in Total Hip Prosthesis. Randomised Study Versus Fixed Insert by Radiostereometric Analysis.
Acronym: DOUMOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08-114
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2015-08

CONDITIONS: Total Hip Replacement
MeSH Terms: interventions — Quartz Crystal Microbalance Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mobility insert with tripod attachment (Novae E®) (Other): mobility insert with tripod attachment (Novae E®)
  Interventions: Device: Novae E®
- mobility insert with press fit pure (Sunfit®) (Other): mobility insert with press fit pure (Sunfit®)
  Interventions: Device: Sunfit®
- fixed insert (Quartz®). (Other): fixed insert (Quartz®).
  Interventions: Device: Quartz®

INTERVENTIONS:
Device: Novae E®
  Arms: mobility insert with tripod attachment (Novae E®)
Device: Sunfit®
  Arms: mobility insert with press fit pure (Sunfit®)
Device: Quartz®
  Arms: fixed insert (Quartz®).

SUMMARY:
The total hip replacement, with over 120,000 cases per year in France, provides short term, excellent functional results and a significant improvement in quality of life, in almost all cases. However, observation showed that the dislocation is not a rare complication (2-4%) and the lifetime of the implants is limited due to aseptic loosening.

The evaluation process used in this study will be the extent of penetration of the metal femoral head in the cup and micro mobility metal back by radiostereometric analysis (RSA) whose precision provides early results (2 3 years), long before wear and migration are measurable by conventional radiological means. The main objective will be to compare, 2 years after the intervention, the penetration of the metal femoral head in 3 types of inserts: two dual mobility inserts, one at tripod attachment (Novae E®), the other press fit pure (Sunfit®), and a fixed insert (Quartz®).

This is a randomized controlled trial. 105 patients will be enrolled (35 in each group). Patients will be included in each of the two participating centers (Amiens, Caen). The analysis will be made in RSA D7 + 2, 6 months 1, 12 months 1 24 months 1. An assessment will be made to 3 years if the analysis requires it to 2 years.

Analysis of pictures will be centralized in Caen and performed with specific software after transferring images via a secure network.

ELIGIBILITY:
Inclusion Criteria:

* patients older men or women 60-75 years
* with a primary or secondary osteoarthritis or osteonecrosis
* having a functional disorder requiring the installation of a total hip prosthesis of primary

Exclusion Criteria:

* patients aged 76 years or more
* protected adults
* resumption of PTH
* cephalic prosthesis recovery or intermediate
* resumption of cupules
* primary or secondary malignant tumor of the hip

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Measuring the penetration of the femoral head in the polyethylene inserts by radiostereometric analysis (RSA) | change over baseline and 3 years